CLINICAL TRIAL: NCT00596570
Title: Management of Patients With Atrial Fibrillation Undergoing Coronary Artery Stenting: A Multicenter, Prospective Registry
Brief Title: Management of Patients With Atrial Fibrillation Undergoing Coronary Artery Stenting
Acronym: AFCAS
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Juhani Airaksinen, University of Turku
Other Study IDs: 12007
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2007-12

CONDITIONS: Atrial Fibrillation; Oral Anticoagulation; Percutaneous Coronary Intervention
Keywords: Atrial fibrillation; Oral Anticoagulation; Percutaneous coronary intervention
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anticoagulation samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patient with atrial fibrillation who underwent PCI
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — Percutaneous coronary interventiom

SUMMARY:
Treatment of patients suffering from atrial fibrillation pose problems when percutaneous coronary intervention with stent implantation (PCI-S) is performed. In the absence of solid evidence-based data, no definite recommendations for the management of this patient subset are currently given in the guidelines on percutaneous coronary intervention issued by the most prominent Cardiology Associations. The management of the antithrombotic treatment before invasive cardiac procedures is also incompletely defined. In this study we aim to determine in patients with atrial fibrillation undergoing PCI-S:

1. the contemporary antithrombotic management;
2. the relative safety and efficacy of the various post-PCI antithrombotic regimens;
3. the safety and efficacy of drug-eluting stents (DES), bare-metal stents (BMS), and bioactive stents (BAS);
4. the safety of various periprocedural antithrombotic strategies including glycoprotein IIb/IIIa inhibitors and bivalirudin;
5. safety and efficacy of radial vs femoral approach.

DETAILED DESCRIPTION:
AFCAS study is an observational, multi-center, prospective registry including patients with atrial fibrillation undergoing PCI-S. Follow-up time is 12 months.

Primary end points are major hemorrhagic and thrombotic/thromboembolic complications including cardiac death and secondary endpoints are Major adverse cardiac events (i.e., need for urgent re-revascularization, myocardial infarction, death), stent thrombosis and major/non major hemorrhagic complications. Clinical follow-up will be completed for all patients via telephone, or clinic visits scheduled at 1, 3, 6, and 12 months after PCI-S. The 1 and 6 months visits are optional. The patients will be asked about their clinical outcomes, hospitalizations and medications. Any additional information needed, such as specific mortality, will be obtained by contacting one of the patient's physicians or other health care professional or from death certificates. CRFs will be completed and faxed without delays after discharge, and after each follow up visit. Recruitment will take approximately 12 months. Follow-up will be 12 months for each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation who undergo PCI.

Exclusion Criteria:

* Because of the observational design, no exclusion criteria are provided.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with atrial fibrillation undergoing PCI-S.
Sampling Method: Probability Sample
Enrollment: 996 (Actual)
Dates: Start 2007-01; Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
major hemorrhagic and thrombotic/thromboembolic complications including cardiac death | one year

CONTACTS AND LOCATIONS:
Overall Officials: Juhani KE Airaksinen, Professor, Principal Investigator — University of Turku
Locations (1):
- Juhani Airaksinen, Turku, Finland

REFERENCES:
- [Derived] Puurunen M, Kiviniemi T, Nammas W, Schlitt A, Rubboli A, Nyman K, Karjalainen P, Kirchhof P, Lip GY, Airaksinen JK. Impact of anaemia on clinical outcome in patients with atrial fibrillation undergoing percutaneous coronary intervention: insights from the AFCAS registry. BMJ Open. 2014 May 13;4(5):e004700. doi: 10.1136/bmjopen-2013-004700. PMID 24823675
- [Derived] Rubboli A, Schlitt A, Kiviniemi T, Biancari F, Karjalainen PP, Valencia J, Laine M, Kirchhof P, Niemela M, Vikman S, Lip GY, Airaksinen KE; AFCAS Study Group. One-year outcome of patients with atrial fibrillation undergoing coronary artery stenting: an analysis of the AFCAS registry. Clin Cardiol. 2014 Jun;37(6):357-64. doi: 10.1002/clc.22254. Epub 2014 Jan 30. PMID 24481953
- [Derived] Schlitt A, Rubboli A, Lip GY, Lahtela H, Valencia J, Karjalainen PP, Weber M, Laine M, Kirchhof P, Niemela M, Vikman S, Buerke M, Airaksinen KE; AFCAS (Management of patients with Atrial Fibrillation undergoing Coronary Artery Stenting Study Group). The management of patients with atrial fibrillation undergoing percutaneous coronary intervention with stent implantation: in-hospital-data from the Atrial Fibrillation undergoing Coronary Artery Stenting study. Catheter Cardiovasc Interv. 2013 Dec 1;82(7):E864-70. doi: 10.1002/ccd.25064. Epub 2013 Aug 28. PMID 23765437